CLINICAL TRIAL: NCT05956457
Title: Evaluating Patient-Reported Outcomes and Wearable Data Among Individuals With Relapsed/Refractory Multiple Myeloma
Brief Title: PRO and Wearable Data Insights From Individuals With R/R Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pack Health (Industry)
Collaborators: University of Washington (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00016359
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma; Relapsed Hematologic Malignancy
Keywords: Digital health; Patient reported outcomes; Wearable Activity Trackers
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: A single cohort of 100 individuals with relapsed/refractory multiple myeloma will be enrolled in the study, all of which will be enrolled in a digital health coaching program and receive a Fitbit device for activity tracking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Cohort Receiving Digital Health Coaching (Experimental): All study participants will be enrolled in a 3-month digital health coaching program. They will also receive a Fitbit device to be worn daily for the capture of physical activity data.
  Interventions: Behavioral: Digital Health Coaching Program; Device: Fitbit

INTERVENTIONS:
Behavioral: Digital Health Coaching Program — Digital health intervention consisting of weekly calls from a Health Advisor to a participant, accompanied by delivery of evidence-based content across health and wellness domains (e.g. nutrition, exercise, physical, emotional and financial health) up to 4 times weekly via text, email or mobile application.
  Other Names: Pack Health Digital Health Coaching
Device: Fitbit — A wrist-worn activity tracker allowing for the capture of physical activity, including but not limited to step-count and minutes of activity, to be captured daily.
  Other Names: Charge 5

SUMMARY:
This study will evaluate the feasibility of a digital health coaching program for adults with relapsed or refractory multiple myeloma (R/R MM). One hundred adults with R/R MM will be enrolled at The University of Washington. Individuals who agree to take part in the study and sign an informed consent will be enrolled in a 3-month digital health coaching program. The program will provide weekly phone calls plus the delivery of learning materials to text or email. Questionnaires and data from a wrist-worn activity tracker will be collected. Outcomes include treatment and symptom experience, quality of life, financial burden, and how confident people feel to manage their health. Information about your condition and treatment will be collected, along with how often you use services like the emergency room, for care. This data will provide a better understanding of how a person experiences their R/R MM.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a chronic malignancy with no current cure. Previously dependent on myeloablative chemotherapy and stem cell transplantation to induce prolonged remission, recent advances in targeted therapies are enhancing overall survival and extending the duration between treatments. Monoclonal antibodies, including CD38-directed monoclonal antibodies, combination immunotherapies, and T-cell therapies are among the many promising agents for treating relapsed or refractory (R/R) MM. This improvement in treatment outcomes is accompanied by significant risk for toxicities such a neutropenia and subsequent infections which themselves can be life-threatening. Several studies indicate a high symptom burden and poor health-related quality of life for individuals with multiple myeloma, with most of what is known from clinical trials of highly selective populations or qualitative studies conducted outside of the US among mostly white patients. These factors, coupled with the rapidly changing multiple myeloma treatment landscape, limits the generalizability to wider population as well as an understanding of MM's impact across the disease course. A more complete investigation of the symptom burden, health self-efficacy, and financial, physiologic, and psychosocial well-being among patients with multiple myeloma is urgently needed to provide a comprehensive view of the ways in which multiple myeloma and its treatments affects individuals' lives.

The purpose of this study is to explore the use of symptom monitoring and digital life coaching (DLC) to inform a more complete understanding of the impact of multiple myeloma on symptom burden, health self-efficacy, and financial, physiologic, and psychosocial well-being among a diverse U.S.-based, contemporary sample. The benefits of routine symptom monitoring have been demonstrated in recent studies, where overall survival increased among cancer patients who routinely monitored their symptoms. As the science related to symptom monitoring continues to evolve, exploring interventions to support both the assessment of and interventions related to disease and treatment-related sequelae it is important to identify how symptoms can best be monitored and managed. Studies to date have explored how symptom monitoring can be conducted for patients in the ambulatory setting, where patients do not receive around the clock assessment and management as they would in the hospital setting. In this context, digital or eHealth technologies are increasingly emerging as ways to promote health behaviors, and to monitor individuals with chronic health states, including cancer. An integrative review of 28 articles specifically evaluating eHealth interventions for patients with cancer identified 16 unique eHealth interventions, largely centered around educational support and decision aids. Telehealth counseling and navigation was found to be effective in supporting psychosocial needs in a small study (n=20) of underserved (defined by the authors as those who were primarily unemployed and uninsured) breast cancer patients. In a study of 1371 cancer patients, 71% reported using a mobile phone daily and 93% reported having internet access from home, of which 68% reported daily internet use, suggesting that internet-based technologies may be purposeful in the sharing of information with and coordination of care for cancer patients. Despite literature indicating its potential efficacy, few interventional studies have been published that evaluate digital health coaching and its relationship with self-efficacy and symptom management, specifically in R/R MM patients. As such, there is a gap in the literature on how digital health coaching might be used to support patients during cancer treatment and into survivorship.

Pack Health, LLC is an independent, patient engagement company that was established in 2014 with the mission of helping patients access the right care for their condition and develop the self-management skills to achieve better health and overall well-being. Pack Health offers a symptom management program involving both interpersonal interactions as well as e-modules for patients diagnosed with cancer to better manage pain, fatigue, depression, anxiety and navigate their care more effectively through digital health coaching and tools.

A recent pilot study at UCSF conducted in collaboration with Pack Health examined the impact of digital life coaching (DLC) on symptom outcomes for individuals with MM undergoing upfront stem cell transplantation. Outcomes suggest the efficacy of a coaching program for engagement up to day +100 post-transplant, with 73% (n=11) DLC engagement and 94% PRO completion. A randomized study of DLC versus usual care in individuals with MM undergoing upfront stem cell transplantation is underway. However, patients with R/R MM (where the disease has come back after prior lines of therapy such as transplantation) may have unique needs. An opportunity exists to explore how a digital health coaching platform might be used for symptom monitoring and coaching during treatment for R/R MM for whom the chronic nature of therapy may influence both needs and outcomes in relation to a DLC intervention.

This is a prospective study of patients with R/R MM to evaluate the feasibility and preliminary outcomes of DLC and its potential to augment existing standards of care for patient support. Patients enrolled in the program will be assigned to a health advisor who will act as an educator and accountability partner, supporting patients as they experience treatment for R/R MM. Throughout the engagement, patient reported outcomes (PROs) will be collected at multiple time points to assess the patient status and will be used to explore relationships between medical management, health related quality of life (HRQoL), and engagement in the program. Patients will be enrolled and will complete all assessments at baseline, 30, 60 and 90 days after consent. Findings from this study will establish feasibility of a DLC intervention for individuals with R/R MM and provide greater insight into their symptom burden, health self-efficacy, and financial, physiologic, and psychosocial well-being through the integration of patient reported, wearable and clinical data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Confirmed diagnosis of MM as determined by participants' primary physicians at the study site. Patients with concurrent AL amyloidosis will be eligible.
3. Initiation of at least the second line of MM-directed therapy for multiple myeloma at time of study enrollment. Participants must have been exposed to at least one proteasome inhibitor (PI) and/or one immunomodulatory drug (IMiD).

Exclusion Criteria:

1. Individuals who are terminally ill, defined as individuals identified by their physician as likely having 6 months or less to live, or those individuals transitioned to comfort measures only (meaning only supportive care measures without curative focused treatment)
2. Individuals who have previously participated in Pack Health digital health coaching
3. Physician-assessed lack of sufficient English proficiency
4. Lack of ownership of a personal smartphone or device allowing for access to text, email or mobile application
5. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with participant's safety, provision of informed consent, or compliance with study procedures
6. Concurrent enrollment on a therapeutic study in R/R MM that precludes simultaneous enrollment onto our non-therapeutic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Digital Health Coaching Intervention | At 3 months following the start of the coaching intervention
  A retention rate greater than or equal to 70%. Retention is defined as individuals who agree to participate in the digital health coaching program and complete the 3 months of engagement post-enrollment. Engagement is defined as the completion of 1 nudge (call, text, or email) per module out of 5 nudge opportunities

SECONDARY OUTCOMES:
Change in Cancer Behavior Inventory-Brief Form (CBI-B) | Change in baseline perception of treatment experience at 3 months
  This 12-item instrument measures self-efficacy in coping with cancer across 7 domains. These include: Seeking and Understanding Medical Information, Emotion Regulation, Coping with Treatment Related Side Effects, Accepting Cancer/ Maintaining a Positive Attitude, Seeking Social Support, and Using Spiritual Coping. The instrument utilizes a 9-point response scale ranging from 1 "Not at all confident" to 9 "Confident".

OTHER OUTCOMES:
Change in Center for Adherence Support Evaluation (CASE) Medication Adherence Index | Change in baseline perception of treatment experience at 3 months
  The Center for Adherence Support Evaluation (CASE) is a three-item questionnaire used to measure antiretroviral therapy adherence. This questionnaire was developed through the Special Projects of National Significance (SPNS) initiative called Assessing Existing Efforts to Increase Adherence to Medication. Patients take less than 5 minutes to answer the three unique questions, asking about their difficulty taking medications on time, average days per week with one dose missed, and the last time they missed a dose.
Change in Comprehensive Score for Financial Toxicity (COST) Instrument | Change in baseline perception of treatment experience at 3 months
  The Comprehensive Score for Financial Toxicity (COST) is an 11-item instrument used to measure the financial toxicity of cancer treatment, which has been demonstrated to be highly correlated with HRQoL (de Souza et al., 2017). This instrument was validated among individuals with advanced cancer and demonstrated high internal consistency (Cronbach's α >.90) and highly correlated to HRQol (p=.05). The instrument consists of 11 items, utilizing a five-point ordinal scale ranging from (0- Not at all) to (4- Very much).
Change in Patient Health Questionnaire (PHQ) 4 | Change in baseline perception of treatment experience at 3 months
  The Patient Health Questionnaire-4 (PHQ-4) is a 4-item inventory rated on a 4-point Likert-type scale. Its items are drawn from the first two items of the 'Generalized Anxiety Disorder-7 scale' (GAD-7) and the 'Patient Health Questionnaire-8' (PHQ-8). Its purpose is to allow for very brief and accurate measurement of depression and anxiety.
Change in Patient Reported Outcomes (PRO)-Common Terminology for Clinically Adverse Events (CTCAE) Blurry Vision Severity and Interference items | Change in baseline perception of treatment experience at 3 months
  The PRO-CTCAE is a validated bank of 124 items representing patient experience of frequency, severity, interference, amount, and presence/absence of 78 symptomatic toxicities from the CTCAE. Responses are scored from 0 (absent) to 4 (severe/very much). We will administer 2 PRO-CTCAE instruments for: severity and interference of blurred vision.
Physical Activity | From date of enrollment up to 3 months
  Minutes of physical activity will be collected via Fitbits provided to study participants
Physical Activity | From date of enrollment up to 3 months
  Daily step count will be collected via Fitbits provided to study participants
Digital Engagement | From date of enrollment up to 3 months
  Duration of engagement with the digital health coaching platform
Digital Engagement | From date of enrollment up to 3 months
  Frequency of engagement with the digital health coaching platform
Digital Engagement | From date of enrollment up to 3 months
  Methods of engagement with the digital health coaching platform

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Cocks K, Cohen D, Wisloff F, Sezer O, Lee S, Hippe E, Gimsing P, Turesson I, Hajek R, Smith A, Graham L, Phillips A, Stead M, Velikova G, Brown J; EORTC Quality of Life Group. An international field study of the reliability and validity of a disease-specific questionnaire module (the QLQ-MY20) in assessing the quality of life of patients with multiple myeloma. Eur J Cancer. 2007 Jul;43(11):1670-8. doi: 10.1016/j.ejca.2007.04.022. Epub 2007 Jun 15. PMID 17574838
- [Background] Cormican O, Dowling M. Managing relapsed myeloma: The views of patients, nurses and doctors. Eur J Oncol Nurs. 2016 Aug;23:51-8. doi: 10.1016/j.ejon.2016.04.003. Epub 2016 May 11. PMID 27456375
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Girault A, Ferrua M, Lalloue B, Sicotte C, Fourcade A, Yatim F, Hebert G, Di Palma M, Minvielle E. Internet-based technologies to improve cancer care coordination: current use and attitudes among cancer patients. Eur J Cancer. 2015 Mar;51(4):551-557. doi: 10.1016/j.ejca.2014.12.001. Epub 2015 Feb 4. PMID 25661828
- [Background] Hari P. Recent advances in understanding multiple myeloma. Hematol Oncol Stem Cell Ther. 2017 Dec;10(4):267-271. doi: 10.1016/j.hemonc.2017.05.005. Epub 2017 Jun 13. PMID 28633036
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Heitzmann CA, Merluzzi TV, Jean-Pierre P, Roscoe JA, Kirsh KL, Passik SD. Assessing self-efficacy for coping with cancer: development and psychometric analysis of the brief version of the Cancer Behavior Inventory (CBI-B). Psychooncology. 2011 Mar;20(3):302-12. doi: 10.1002/pon.1735. PMID 20878830
- [Background] Kelly M, Dowling M. Patients' lived experience of myeloma. Nurs Stand. 2011 Mar 16-22;25(28):38-44. doi: 10.7748/ns2011.03.25.28.38.c8397. PMID 21488448
- [Background] Kent EE, Ambs A, Mitchell SA, Clauser SB, Smith AW, Hays RD. Health-related quality of life in older adult survivors of selected cancers: data from the SEER-MHOS linkage. Cancer. 2015 Mar 1;121(5):758-65. doi: 10.1002/cncr.29119. Epub 2014 Nov 4. PMID 25369293
- [Background] LeBlanc MR, Hirschey R, Leak Bryant A, LeBlanc TW, Smith SK. How are patient-reported outcomes and symptoms being measured in adults with relapsed/refractory multiple myeloma? A systematic review. Qual Life Res. 2020 Jun;29(6):1419-1431. doi: 10.1007/s11136-019-02392-6. Epub 2019 Dec 17. PMID 31848847
- [Background] Lee MK, Schalet BD, Cella D, Yost KJ, Dueck AC, Novotny PJ, Sloan JA. Establishing a common metric for patient-reported outcomes in cancer patients: linking patient reported outcomes measurement information system (PROMIS), numerical rating scale, and patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Patient Rep Outcomes. 2020 Dec 10;4(1):106. doi: 10.1186/s41687-020-00271-0. PMID 33305344
- [Background] Lowe B, Wahl I, Rose M, Spitzer C, Glaesmer H, Wingenfeld K, Schneider A, Brahler E. A 4-item measure of depression and anxiety: validation and standardization of the Patient Health Questionnaire-4 (PHQ-4) in the general population. J Affect Disord. 2010 Apr;122(1-2):86-95. doi: 10.1016/j.jad.2009.06.019. Epub 2009 Jul 17. PMID 19616305
- [Background] Madduri D, Dhodapkar MV, Lonial S, Jagannath S, Cho HJ. SOHO State of the Art Updates and Next Questions: T-Cell-Directed Immune Therapies for Multiple Myeloma: Chimeric Antigen Receptor-Modified T Cells and Bispecific T-Cell-Engaging Agents. Clin Lymphoma Myeloma Leuk. 2019 Sep;19(9):537-544. doi: 10.1016/j.clml.2019.08.002. Epub 2019 Aug 7. PMID 31427259
- [Background] Madore S, Kilbourn K, Valverde P, Borrayo E, Raich P. Feasibility of a psychosocial and patient navigation intervention to improve access to treatment among underserved breast cancer patients. Support Care Cancer. 2014 Aug;22(8):2085-93. doi: 10.1007/s00520-014-2176-5. Epub 2014 Mar 18. PMID 24639035
- [Background] Maher K, de Vries K. An exploration of the lived experiences of individuals with relapsed multiple myeloma. Eur J Cancer Care (Engl). 2011 Mar;20(2):267-75. doi: 10.1111/j.1365-2354.2010.01234.x. Epub 2010 Oct 18. PMID 20950368
- [Background] Mannheimer SB, Mukherjee R, Hirschhorn LR, Dougherty J, Celano SA, Ciccarone D, Graham KK, Mantell JE, Mundy LM, Eldred L, Botsko M, Finkelstein R. The CASE adherence index: A novel method for measuring adherence to antiretroviral therapy. AIDS Care. 2006 Oct;18(7):853-61. doi: 10.1080/09540120500465160. PMID 16971298
- [Background] Moreno L, Perez C, Zabaleta A, Manrique I, Alignani D, Ajona D, Blanco L, Lasa M, Maiso P, Rodriguez I, Garate S, Jelinek T, Segura V, Moreno C, Merino J, Rodriguez-Otero P, Panizo C, Prosper F, San-Miguel JF, Paiva B. The Mechanism of Action of the Anti-CD38 Monoclonal Antibody Isatuximab in Multiple Myeloma. Clin Cancer Res. 2019 May 15;25(10):3176-3187. doi: 10.1158/1078-0432.CCR-18-1597. Epub 2019 Jan 28. PMID 30692097
- [Background] Nielsen LK, Jarden M, Andersen CL, Frederiksen H, Abildgaard N. A systematic review of health-related quality of life in longitudinal studies of myeloma patients. Eur J Haematol. 2017 Jul;99(1):3-17. doi: 10.1111/ejh.12882. Epub 2017 Apr 25. PMID 28322018
- [Background] Osoba D, Aaronson N, Zee B, Sprangers M, te Velde A. Modification of the EORTC QLQ-C30 (version 2.0) based on content validity and reliability testing in large samples of patients with cancer. The Study Group on Quality of Life of the EORTC and the Symptom Control and Quality of Life Committees of the NCI of Canada Clinical Trials Group. Qual Life Res. 1997 Mar;6(2):103-8. doi: 10.1023/a:1026429831234. PMID 9161109
- [Background] Proskorovsky I, Lewis P, Williams CD, Jordan K, Kyriakou C, Ishak J, Davies FE. Mapping EORTC QLQ-C30 and QLQ-MY20 to EQ-5D in patients with multiple myeloma. Health Qual Life Outcomes. 2014 Mar 11;12:35. doi: 10.1186/1477-7525-12-35. PMID 24618388
- [Background] Ramsenthaler C, Kane P, Gao W, Siegert RJ, Edmonds PM, Schey SA, Higginson IJ. Prevalence of symptoms in patients with multiple myeloma: a systematic review and meta-analysis. Eur J Haematol. 2016 Nov;97(5):416-429. doi: 10.1111/ejh.12790. Epub 2016 Sep 6. PMID 27528496
- [Background] Rothwell PM. External validity of randomised controlled trials: "to whom do the results of this trial apply?". Lancet. 2005 Jan 1-7;365(9453):82-93. doi: 10.1016/S0140-6736(04)17670-8. PMID 15639683
- [Background] Schumacher A, Kessler T, Buchner T, Wewers D, van de Loo J. Quality of life in adult patients with acute myeloid leukemia receiving intensive and prolonged chemotherapy -- a longitudinal study. Leukemia. 1998 Apr;12(4):586-92. doi: 10.1038/sj.leu.2400977. PMID 9557618
- [Background] Schumacher A, Wewers D, Heinecke A, Sauerland C, Koch OM, van de Loo J, Buchner T, Berdel WE. Fatigue as an important aspect of quality of life in patients with acute myeloid leukemia. Leuk Res. 2002 Apr;26(4):355-62. doi: 10.1016/s0145-2126(01)00145-x. PMID 11839378
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Ventura F, Ohlen J, Koinberg I. An integrative review of supportive e-health programs in cancer care. Eur J Oncol Nurs. 2013 Aug;17(4):498-507. doi: 10.1016/j.ejon.2012.10.007. Epub 2012 Nov 15. PMID 23158437
- [Background] Zaleta AK, Miller MF, Olson JS, Yuen EYN, LeBlanc TW, Cole CE, McManus S, Buzaglo JS. Symptom Burden, Perceived Control, and Quality of Life Among Patients Living With Multiple Myeloma. J Natl Compr Canc Netw. 2020 Aug;18(8):1087-1095. doi: 10.6004/jnccn.2020.7561. PMID 32755984
- [Background] Zhang T, Wang S, Lin T, Xie J, Zhao L, Liang Z, Li Y, Jiang J. Systematic review and meta-analysis of the efficacy and safety of novel monoclonal antibodies for treatment of relapsed/refractory multiple myeloma. Oncotarget. 2017 May 16;8(20):34001-34017. doi: 10.18632/oncotarget.16987. PMID 28454113
- [Background] Banerjee R, Huang CY, Dunn L, Knoche J, Ryan C, Brassil K, Jackson L, Patel D, Lo M, Arora S, Wong SW, Wolf J, Martin Iii T, Dhruva A, Shah N. Digital Life Coaching During Stem Cell Transplantation: Development and Usability Study. JMIR Form Res. 2022 Mar 4;6(3):e33701. doi: 10.2196/33701. PMID 35039279